CLINICAL TRIAL: NCT00835029
Title: Efficacy of Slow Release Clotrimazole Varnish Treating Denture Stomatitis
Brief Title: Efficacy of Slow Release Clotrimazole Varnish Treating Denture Stomatitis Comparing to Traditional Treatment of Troches
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Czerninski Rakefet, Dr, Oral diseases clinic, Hadassah Medical Organization
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111111
Record Dates: First submitted 2009-02-01; First posted 2009-02-03 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 2015-03

CONDITIONS: Oral Candidiasis; Denture Stomatitis
Keywords: oral; candida; denture; clotrimazole; slow releases
MeSH Terms: conditions — Candidiasis, Oral; Stomatitis, Denture; Torulopsis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clotrimazole varnish (Active Comparator): Clotrimazole in a slow release varnish treatment
  Interventions: Drug: Clotrimazole varnish
- Clotrimazole troches (Active Comparator): Clotrimazole troches 10 mgx5 day for treatment of denture associated candiad infection
  Interventions: Drug: Clotrimazole troches

INTERVENTIONS:
Drug: Clotrimazole varnish — Each patient will receive 14 syringes (with no needle, equivalent to 50 mg of Clotrimazole in each one) . The varnish will be applied on a dried denture at the inner side by means of a soft brush and left to dry for 60 sec for 14 days.
  Other Names: Oralten
  Arms: Clotrimazole varnish
Drug: Clotrimazole troches — The troche group will be asked to dissolve it in the mouth according to the manufacture instructions five times a day after removal of the denture, for 14 days.
  Other Names: Oralten
  Arms: Clotrimazole troches

SUMMARY:
Background: Oral candidiasis is most frequently found among the elderly .It is accompanied with oral pain, irritation, burning sensation. In addition, the altered taste sensation may cause nutrition compromise, which may affect ones diet. Management of superficial oral Candida is usually achieved by treatment with clotrimazole, a fungi static drug which is given five times per day with instruction to slowly suck on it with out the dentures.

Working hypothesis and aims: Management of oral candidiasis is feasible. The major disadvantage of the mode of action now days is the substantively of the drug in the oral cavity and patient compliance. A sustained release varnish which is easily applied on the dentures, which also release the anti fungal drug for at least a day, may overcome some of the pit falls of the treatment applied today.

Based on our past experience, in developing local sustained release varnishes for dental use, we anticipate that we can also formulate a special anti fungal sustained release varnish which will fit the special and unique needs of the elderly population.

Methods: Sustained release varnish will be developed in our laboratory. The kinetics of release (using HPLC) and antifungal activity (Bioassays) will be examined in vitro. The formulation showing the optimal results will be tested on human subjects with oral candidiasis. The efficacy of the varnish will be examined clinically (reduction in symptoms), microbiology (reduction of oral fungal), pharmaceutically (release kinetics in vivo).

Expected results: The clinical out come of one time varnish application will be improved compared to the five times application of lozenges (used today). The severity of the disease should decrease and the healing period should be shorten drastically.

Importance: This is a novel pharmaceutical development of a local application of a dental varnish designed specially to the elderly population

ELIGIBILITY:
Inclusion Criteria:

* adults
* removable denture in mouth
* diagnosed oral candida

Exclusion Criteria:

* allergy to clotrimazole
* immunosuppressed
* using other antifungi treatment
* have an active oral ulcerative disease
* impaired kidny or live functions

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Microbial evidence of reduced candida infection | one and two weeks after inevention

SECONDARY OUTCOMES:
Clinical evidence for candida infection | One and two weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rakefet Czerninski, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hdassah medical Organization,, Jerusalem, Israel